CLINICAL TRIAL: NCT05757219
Title: A Phase 2, Single-Arm, Open-Label Study Using Itacitinib as Pre-Modulation in Patients With Diffuse Large B-Cell Lymphoma (DLBCL) Receiving CAR-T-Cell Therapy
Brief Title: Itacitinib Pre-modulation in DLBCL Receiving CAR T Cell Therapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-21892
Record Dates: First submitted 2023-02-24; First posted 2023-03-07 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Diffuse Large B Cell Lymphoma
Keywords: CAR-T; chimeric antigen receptor (CAR) T-cell therapy
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — itacitinib; Receptors, Chimeric Antigen; Automobiles; axicabtagene ciloleucel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pre-Modulation Treatment (Experimental): Participants will receive itacitinib 200 mg PO QD beginning at time of apheresis approximately 4-6 weeks prior to CAR-T-cell therapy and will continue until Day 30 (30 Days Post-CAR-T-cell therapy)
  Interventions: Drug: Itacitinib; Biological: Chimeric antigen receptor (CAR) T-cell therapy

INTERVENTIONS:
Drug: Itacitinib — Participants start itacitinib 200 mg PO once daily within 1-4 days after apheresis while awaiting CAR-T-cell manufacturing, which is expected to take approximately from week -4 until day -7. Patients will remain on itacitinib 200 mg PO once daily from initiation until 30 days post-CAR-T-cell therapy (Day 30) including throughout lymphodepleting chemotherapy period (Days -5, -4, -3) and axi-cel infusion (Day 0) for a total of approximately 58 doses.
Biological: Chimeric antigen receptor (CAR) T-cell therapy — Yescarta is an autologous anti-CD19 CAR T cell therapy manufactured from the patient's own T cells, which have been extracted and then reprogrammed with CAR molecules to help the T cells recognize cancer cells. The reengineered T cells are infused back into the patient to attack the cancer.
  Other Names: YESCARTA; Axi-cel

SUMMARY:
The purpose of the study is to assess the safety and efficacy of once daily itacitinib oral administration in participants with diffuse large B-cell lymphoma (DLBCL) who will receive CAR-T cell therapy with axicabtagene ciloleucel (axi-cel).

DETAILED DESCRIPTION:
This is a phase 2, single-arm, open-label study to assess the safety and efficacy of once daily itacitinib oral administration in patients with diffuse large B-Cell lymphoma (DLBCL) who will receive CAR-T-cell therapy with axicabtagene ciloleucel (Axi-cel) and have been found to have high levels of systemic inflammation. Approximately n=27 adult males and females, 18 years or older, who will receive treatment for diffuse large B-cell lymphoma (DLBCL) at the Moffitt Cancer Center with a ferritin level greater than 400 ng/ml and C-reactive protein (CRP) level greater than 2 mg/dl (20 mg/l) at screening will be enrolled. Study regimen will consist of itacitinib 200 mg PO QD beginning at time of apheresis approximately 4-6 weeks prior to CAR-T-cell therapy and will continue until Day 30 (30 Days Post-CAR-T-cell therapy). The exact number of days between apheresis and CAR T cell infusion may vary based on CAR T cell manufacturing turnaround. A single infusion of axi-cel therapy will be administered on Day 0. Investigators hypothesize that pre-modulation with itacitinib started approximately 4 weeks prior to CAR-T-cell therapy with axi-cel will improve patient outcomes in those patients with diffuse large B-cell lymphoma (DLBCL) who express high levels of systemic inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a histologically confirmed diagnosis of diffuse large B-cell lymphoma (DLBCL) who plan to receive treatment at the Moffitt Cancer Center/
* Adult males or females who are 18 years of age or older at time of signing informed consent.
* Must have ability to comprehend and the willingness to sign written informed consent for study participation.
* Eligible to receive CAR-T cell therapy (axicabtagene ciloleucel) for DLBCL and histological variants.
* Patients must have a serum ferritin level above 400 mg/mL and C-reactive protein level above 2 mg/dL (20 mg/L) at screening.
* ECOG performance status 0 to 2.
* The effects of Itacitinib on the developing human fetus are unknown. For this reason and because Janus kinase (JAK)1-selective inhibitors as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation as outlined in criteria below: (a) Men must agree to take appropriate precautions to avoid fathering children (with at least 99% certainty) from screening through safety follow up and must refrain from donating sperm during this period. Permitted methods that are at least 99% effective in preventing pregnancy should be communicated to the participants in their understanding confirmed.(b) Women of childbearing potential must have a negative serum pregnancy test at screening and before the first dose of Day 1 and must agree to take appropriate precautions to avoid pregnancy (with at least 99% certainty) from screening through safety follow up. Permitted methods that are at least 99% effective in preventing pregnancy should be communicated to the participants and their understanding confirmed. (c) Women of non-childbearing potential (ie, surgically sterile with a hysterectomy and/or bilateral oophorectomy OR >= 12 months of amenorrhea) are eligible.
* Patients must be ineligible for stem cell transplant at screening on the basis of active lymphoma.
* Patients must meet laboratory parameters at screening as defined in protocol

Exclusion Criteria:

* Patients who are currently receiving or who have received any investigational study agent ≤4 weeks prior to screening visit are ineligible.
* Prior treatment with chimeric antigen receptor (CAR) T-cell therapy.
* Participants with clinically significant or uncontrolled cardiac disease, including unstable angina, acute myocardial infarction within 6 months from screening, New York Health Association III or IV heart failure, and circulatory collapse requiring vasopressor or inotropic support
* Participants with arrhythmias that are not stable on a medical management program within 2 weeks of screening are also excluded.
* Participants with arrhythmias that are not stable on a medical management program within 2 weeks of screening are also excluded.
* Evidence of active uncontrolled/untreated infection (viral, bacterial, fungal, opportunistic) of any origin.
* Participants with a known history or prior diagnosis of immunologic or inflammatory/autoimmune disease affecting the CNS, and unrelated to their disease under study or previous treatment.
* Known positive Human immunodeficiency virus (HIV) status.
* Participants with evidence of active and/or chronic hepatitis B virus (HBV) infection, HBV viral load must be undetectable on suppressive therapy, if indicated.
* Participants with a history of hepatitis C virus (HCV) infection, HCV must have been treated and cured.
* Participants who require the concurrent use of chronic systemic steroids or immunosuppressant medications. Steroids should not be given within 5 days prior to leukapheresis. Concomitant bridging steroids (section 6.6) are allowed after leukapheresis.
* Known hypersensitivity or severe reaction to itacitinib, similar compounds, or excipients or itacitinib.
* Participants who have not recovered from adverse events (AEs) due to prior anti-cancer therapy (i.e., have residual toxicities > Grade 1), with the exception of stable Grade 2 peripheral neuropathy and/or any grade alopecia.
* Pregnant or nursing (breast-feeding) women are excluded from this study because there is an unknown but potential risk to using itacitinib in pregnant or nursing women.
* Any condition that would, in the investigator's judgement, interfere with full participation in the study, including administration of itacitinib and attending required study visits (if outpatient); pose a significant risk to the participant; or interfere with interpretation of study data.
* Inability of the participant to swallow and retain oral medication.
* Participants receiving any medications or substances that are strong inhibitors of CYP3A4 are ineligible. As part of the enrollment/informed consent procedures, the participant will be counseled on the risk of interactions with other agents and what to do if new medications need to be prescribed or if the participant is considering a new over-the-counter medicine or herbal product.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2023-05-19 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | at 6 months
  Progression Free Survival is defined as the time from start of treatment to the time of disease progression or death. Among patients treated with axi-cel who have a ferritin >400 ng/ml and CRP>2 mg/dl at the time of apheresis, the 6 month PFS was 25%. The primary endpoint of this study will be met if pre-modulation with itacitinib followed by axi-cel leads to a 6 month PFS of 45% or higher.

SECONDARY OUTCOMES:
Incidence of Severe Cytokine Release Syndrome (CRS) | Up to 3 months
  Number of participants who experience severe (grade 3 or higher by ASTCT criteria) CRS in the first 30 days after CAR-T infusion.
Incidence of Severe Immune efflector cell Associated Neurotoxicity Syndrome (ICANS) | Up to 3 months
  Number of participants who experience severe (grade 3 or higher by ASTCT criteria) ICANS in the first 30 days after CAR-T infusion per CTCAE 5.0.
Overall Response Rate | at 6 months
  Overall Response Rate is defined as the rate of the best overall response as complete response (CR) or partial response (PR) by Lugano Response Criteria. Lugano Criteria are based on PET or bidimensional tumor measurements on computerized tomography (CT).
Overall Survival (OS) | up to 27months
  Overall Survival (OS) will be measured from the initial date of treatment to the recorded date of death.
Progression Free Survival (PFS) | up to 27 months
  Progression Free Survival is defined as the time from start of treatment to the time of disease progression or death. Among patients treated with axi-cel who have a ferritin >400 ng/ml and CRP>2 mg/dl at the time of apheresis, the 6 month PFS was 25%. The primary endpoint of this study will be met if pre-modulation with itacitinib followed by axi-cel leads to a 6 month PFS of 45% or higher.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Jain, MD, PhD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No